CLINICAL TRIAL: NCT02017691
Title: Cerebral Regional Tissue Oxygen Saturation to Guide Oxygen Delivery in Preterm Neonates During Immediate Transition After Birth (COSGOD) - a Prospective Two-centre Randomized Controlled Pilot Feasibility Study
Brief Title: Cerebral Oxygenation to Guide Supplemental Oxygen
Acronym: COSGOD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Pichler Gerhard, MD., Assoc. Prof., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-295
Record Dates: First submitted 2013-11-28; First posted 2013-12-23 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Oxygen Saturation
MeSH Terms: interventions — Spectroscopy, Near-Infrared; Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Near Infrared Spectroscopy (Experimental): crSO2 measurements in addition SpO2 measurements will be visible to guide supplemental oxygen support and respiratory support according predefined interventions depending on the infants breathing efforts and the heart rate during the first 15 minutes after birth
  Interventions: Device: Near Infrared Spectroscopy
- Pulse-oximetry (Other): Only SpO2 measurements will be visible to guide supplemental oxygen support and respiratory support according predefined interventions depending on the infants breathing efforts and the heart rate during the first 15 minutes after birth
  Interventions: Device: Pulse-oximetry

INTERVENTIONS:
Device: Near Infrared Spectroscopy — If crSO2 is <10th centile, CPAP via face mask will be started or oxygen support will be increased depending SpO2, on the infants breathing efforts and the heart rate. If crSO2 remains stable >10th centile, or if crSO2 is > 90th centile CPAP via face mask will be stopped or FiO2 will be reduced depending on SpO2, the infants breathing efforts and the heart rate.
  Arms: Near Infrared Spectroscopy
Device: Pulse-oximetry — If SpO2 remains <10th centile, respiratory support via face mask will be started or FiO2 will be increased depending on the infants breathing efforts and the heart rate. If SpO2 remains stable or if SpO2 is >90th centile respiratory support via face mask will be stopped or FiO2 will be reduced depending on the infants breathing efforts and the heart rate.
  Arms: Pulse-oximetry

SUMMARY:
Objective: Objective of this pilot feasibility study is to monitor crSO2 using NIRS INVOS 5100 (Somanetics, USA) in addition to SpO2 monitoring to guide supplemental oxygen delivery and respiratory support based on both measurements in preterm neonates during the first 15 minutes after birth.

Patients: Preterm neonates <34+0 weeks of gestation born via caesarean section and/or who require respiratory support will be eligible for the study.

Design: A prospective two-centre randomized controlled pilot feasibility study

Methods: Study group: Pulse oximetry will be used to measure SpO2 and heart rate as routine non-invasive monitoring in the first minutes of resuscitation. In addition during the first 15 minutes NIRS measurements will be recorded. crSO2 measurements in addition SpO2 measurements will be used to guide supplemental oxygen support and respiratory support during the first 15 minutes after birth. Control group: Only SpO2 measurements will be used to guide supplemental oxygen support and respiratory support during the first 15 minutes after birth.

Hypothesis: Supplemental oxygen support and respiratory support guided by crSO2 and SpO2 measurements will reduce the time in % minutes of crSO2 <10th or >90th centile in preterm neonates during the first 15 minutes after birth

Outcome Parameter: Primary outcome parameter will be duration in % minute of crSO2 <10th or >90th centile.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonate <34+0 weeks after caesarean section
* Decision to conduct full life support
* Written informed consent

Exclusion Criteria:

* No decision to conduct full life support
* No written informed consent
* Congenital malformation

Max Age: 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cerebral tissue oxygen saturation (crSO2) | 15 minutes
  Duration in % minute of crSO2 <10th or >90th centile

SECONDARY OUTCOMES:
Mortality | 16 weeks
  Rate of mortality
Cerebral injury | 16 weeks
  Cerebral injury assessed by sonography
Neurodevelopmental outcome | 16 weeks
  General movements

OTHER OUTCOMES:
Morbidity | 16 weeks
  Severe morbidities, Rate of intubation during resuscitation, Need of mechanical ventilation on the first day of life,
  Monitoring parameters during the first 15minutes after birth:
  Mean (SD) HR, Mean (SD) BP, Mean (SD) SpO2, NIRS parameters

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, MD, Principal Investigator — Dep. of Pediatrics, Medical University of Graz
Locations (2):
- Department of Pediatrics, Medical University of Graz, Graz, Styria, Austria
- Department of Pediatrics, Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Pichler G, Urlesberger B, Baik N, Schwaberger B, Binder-Heschl C, Avian A, Pansy J, Cheung PY, Schmolzer GM. Cerebral Oxygen Saturation to Guide Oxygen Delivery in Preterm Neonates for the Immediate Transition after Birth: A 2-Center Randomized Controlled Pilot Feasibility Trial. J Pediatr. 2016 Mar;170:73-8.e1-4. doi: 10.1016/j.jpeds.2015.11.053. Epub 2015 Dec 30. PMID 26743498